CLINICAL TRIAL: NCT03208660
Title: A Retrospective Multicenter Study to Investigate Dosage, Efficacy, and Safety of Fycompa in Routine Clinical Care of Patients With Epilepsy
Brief Title: Study to Investigate Dosage, Efficacy, and Safety of Fycompa in Routine Clinical Care of Patients With Epilepsy
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2007-G000-506
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Epilepsy
Keywords: seizure; Fycompa
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fycompa: Participants diagnosed with epilepsy and treated with Fycompa
  Interventions: Drug: Fycompa

INTERVENTIONS:
Drug: Fycompa — Oral suspension
  Other Names: Perampanel

SUMMARY:
This study is conducted to assess the retention rate of Fycompa when given in routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have met all of the following criteria to be included in this study:

  1. Diagnosis of epilepsy
  2. Initiated treatment with Fycompa at any time after 01 Jan 2014
  3. Provided written informed consent by the participant or the participant's legally authorized representative signed for the use of medical records (if required by an Institutional Review Board [IRB] or Independent Ethics Committee [IEC], or by regulatory authorities).

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be obtained by reviewing the medical records of the participants with a diagnosis of epilepsy and treated with Fycompa on clinician's recommendation at up to approximately 40 epilepsy centers.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage of participants remaining on Fycompa treatment at specified time points after initiation of treatment (Retention rate) | 3, 6, 12, 18, and 24 months
  Retention rate is the ratio of the number of participants remaining on Fycompa treatment to the number of participants who could have been exposed for that length of time.

SECONDARY OUTCOMES:
Number of participants with a 50% response rate | up to 24 months
  The response rate will be evaluated from seizure frequencies recorded in medical records or seizure diaries, where available. If not available, the investigator assessment of the therapeutic response will be used.
Number of participants with a 75% response rate | up to 24 months
  The response rate will be evaluated from seizure frequencies recorded in medical records or seizure diaries, where available. If not available, the investigator assessment of the therapeutic response will be used.
Number of participants with a 100% response rate | up to 24 months
  The response rate will be evaluated from seizure frequencies recorded in medical records or seizure diaries, where available. If not available, the investigator assessment of the therapeutic response will be used.
Categorized percent reduction in seizure frequency from baseline | Baseline, up to 24 months
  An epileptic seizure or seizure is a brief episode of signs or symptoms due to abnormal excessive or synchronous neuronal activity in the brain. The outward effect can vary from uncontrolled jerking movement (tonic-clonic seizure) to as subtle as a momentary loss of awareness (absence seizure).
Median percent change in seizure frequency from baseline | Baseline, up to 24 months
  An epileptic seizure or seizure is a brief episode of signs or symptoms due to abnormal excessive or synchronous neuronal activity in the brain. The outward effect can vary from uncontrolled jerking movement (tonic-clonic seizure) to as subtle as a momentary loss of awareness (absence seizure).
Percentage of participants who had no change or a worsening of seizures from baseline | Baseline, up to 24 months
  An epileptic seizure or seizure is a brief episode of signs or symptoms due to abnormal excessive or synchronous neuronal activity in the brain. The outward effect can vary from uncontrolled jerking movement (tonic-clonic seizure) to as subtle as a momentary loss of awareness (absence seizure).
Total provider health care visits before, during, and after final dose of Fycompa | 6 months before initiation of Fycompa to 6 months after last dose of Fycompa
  Total provider health care visits before, during, and after final dose of Fycompa will be summarized as a safety variable.
Number of participants with any treatment-emergent (TE) serious adverse event (SAE) resulting in discontinuation of Fycompa | Up to 24 months
  An SAE is any untoward medical occurrence that at any dose: results in death; is life threatening (ie, the participant was at immediate risk of death from the adverse events [AE] as it occurred; this does not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). A TEAE is defined as an AE that emerges during treatment, having been absent at pretreatment (baseline) or (1) reemerges during treatment, having been present at pretreatment (baseline) but stopped before treatment, or (2) worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Number of participants with any treatment-emergent adverse event (TEAE) resulting in discontinuation of Fycompa | Up to 24 months
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product. A TEAE is defined as an AE that emerges during treatment, having been absent at pretreatment (baseline) or (1) reemerges during treatment, having been present at pretreatment (baseline) but stopped before treatment, or (2) worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Mean change in body weight from baseline | Baseline, Up to 24 months
  Change from baseline is calculated as the post-baseline value minus the baseline value.
Mean change in height of pediatric participants from baseline | Baseline, Up to 24 months
  Change from baseline is calculated as the post-baseline value minus the baseline value.
Maximum dose of Fycompa | Up to 24 months
  The extent of exposure of Fycompa will be determined by summarizing the maximum dose of the study drug.
Average dose of Fycompa | Up to 24 months
  The extent of exposure of Fycompa will be determined by summarizing the average dose of the study drug.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Arizona Age Reversal & Neurology Clinic, Phoenix, Arizona
  - Bronislava Shafran, MD, PC, Phoenix, Arizona
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Arizona Neurological Institute, Sun City, Arizona
  - The University of Arizona Department of Neurology, Tucson, Arizona
  - Valley Children's Hospital, Madera, California
  - UC Davis Medical Center, Sacramento, California
  - Sutter Health, Sacramento, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Capernaum Medical Center, Lakeland, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Pediatric Neurology PA, Orlando, Florida
  - Doctors hospital of Sarasota, Sarasota, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Consultants in Epilepsy & Neurology PLLC, Boise, Idaho
  - Carle Foundation Hospital, Urbana, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health System, Detroit, Michigan
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, Hartsdale, New York
  - Albert Einstein College of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Northwell Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania, Pittsburgh, Pennsylvania
  - Le Bonheur Children's Hospital - PIN, Memphis, Tennessee
  - Austin Epilepsy Center, Austin, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Auburn Neurological Institute, Auburn, Washington
  - Northwest Neurology & Electrodiagnostic Center, Auburn, Washington
  - Seattle Children's Hospital - PIN, Seattle, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington

REFERENCES:
- [Derived] Segal E, Wheless J, Moretz K, Penovich P, Patten A, Malhotra M. Perampanel in real-world clinical care of adolescent and adult patients with epilepsy: Results from the retrospective Phase IV PROVE Study. Seizure. 2022 May;98:87-94. doi: 10.1016/j.seizure.2022.02.011. Epub 2022 Feb 26. PMID 35453064
- [Derived] Segal E, Moretz K, Wheless J, Penovich P, Lancman M, Patten A, Malhotra M. PROVE-Phase IV Study of Perampanel in Real-World Clinical Care of Patients with Epilepsy: Interim Analysis in Pediatric Patients. J Child Neurol. 2022 Mar;37(4):256-267. doi: 10.1177/08830738211047665. Epub 2022 Jan 7. PMID 34994582
- [Derived] Wechsler RT, Wheless J, Zafar M, Huesmann GR, Lancman M, Segal E, Chez M, Aboumatar S, Patten A, Salah A, Malhotra M. PROVE: Retrospective, non-interventional, Phase IV study of perampanel in real-world clinical care of patients with epilepsy. Epilepsia Open. 2022 Jun;7(2):293-305. doi: 10.1002/epi4.12575. Epub 2022 Mar 20. PMID 34942053
- [Derived] Wheless J, Wechsler RT, Lancman M, Aboumatar S, Patten A, Malhotra M. Perampanel in real-world clinical care of patients with epilepsy: Interim analysis of a phase IV study. Epilepsia Open. 2020 Dec 19;6(1):79-89. doi: 10.1002/epi4.12445. eCollection 2021 Mar. PMID 33681651